CLINICAL TRIAL: NCT03569410
Title: The Effect of Natural Protein vs. Protein Supplements on Peritoneal Dialysis Patients An Open-label Prospective Clinical Trial
Brief Title: The Effect of Natural Protein vs. Protein Supplements on Peritoneal Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11101
Record Dates: First submitted 2018-05-22; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Peritoneal Dialysis Complication; Hypoalbuminemia; Malnutrition
Keywords: peritoneal dialysis; albumin; end stage renal disease
MeSH Terms: conditions — Hypoalbuminemia; Malnutrition; Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Open-label prospective clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement Group (Active Comparator): The protein supplement group was instructed by their dietician in how many protein supplements to consume in addition to their natural food intake in order to reach their goal protein intake.
  Interventions: Behavioral: increase protein intake via protein supplements
- Natural Food Group (Experimental): The Natural food group was instructed by their dietician in how much additional protein rich foods to eat in order to reach their goal protein intake.
  Interventions: Behavioral: increased protein intake via natural foods

INTERVENTIONS:
Behavioral: increased protein intake via natural foods — Patients had to eat 1.4g/kg/day of natural protein.
  Arms: Natural Food Group
Behavioral: increase protein intake via protein supplements — Patients ate enough protein supplements in addition to their regular diet to reach eat 1.4g/kg/day of protein intake.
  Arms: Supplement Group

SUMMARY:
This study is a prospective open label clinical trial comparing serum albumin levels and total protein intake in the peritoneal dialysis patient population. A total of 60 patients were enrolled, 16 chose to be in the natural food group and 44 in the supplement group. 4 were lost to follow-up in the supplement group leading to an n of 40. Both groups were educated by dietitians on how to increase their protein intake to a goal of 1.4g/kg/day. The groups were followed for 3 months with protein intake calculated according to the patient's food diaries. Patient demographics and characteristics were compared in both groups.

DETAILED DESCRIPTION:
This is a prospective open label clinical trial comparing serum albumin levels and total protein intake in the peritoneal dialysis patient population. Two treatment groups were established: a natural food group who was instructed by their dietician in how to reach their goal protein intake through purely increasing the consumption of natural foods rich in protein versus a protein supplement group who was instructed by their dietician in how many protein supplements to consume in addition to their natural food intake in order to reach their goal protein intake. To increase compliance, patients were allowed to choose which treatment group they wanted to participate in. Patients, however, were not allowed to change groups during the study.

At the initiation of the study patients were asked to record food diaries so the dietician can calculate their baseline protein intake. Each patient had an assigned dietician who met with the patient monthly. The food diaries were collected during their monthly visits. Patients were also randomly called and asked to give their food intake during the last 24 hours in order to minimize recall bias. Each month the participant's dietician calculated their protein intake deficit and educated the patient on how to increase their protein intake to reach their goal of 1.4g/kg/day. The recommended protein intake for peritoneal dialysis patients is between 1.2 to 1.5 g/kg/day. Therefore, a goal of 1.4g/kg/day was set, which is at the higher end of the goal range in order to ensure an adequately high protein intake.

The patient's serum albumin levels, phosphate levels, kt/v, and total protein intake were recorded at baseline, month 1 (M1), month 2 (M2), and month 3 (M3). Furthermore, all major comorbidities in each patient were recorded and compared. Data was extracted from the electronical medical record system and entered into a password protected file. This data was then analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Initiation of peritoneal dialysis for at least a one-month time period, with the expectation to stay on peritoneal dialysis for the next 3 months
* Independence with all activities of daily living (especially being able to cook)

Exclusion Criteria:

* Age under 18 years
* Expectation of termination of peritoneal dialysis within 3 months of entering the study
* Life expectancy less than three months
* Termination of life or peritoneal dialysis during the study period
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Serum Albumin Levels | After three months of intervention.
  serum levels of albumin

SECONDARY OUTCOMES:
Serum Phosphorus levels | At Month 0, 1, 2, and 3
  measured monthly
Goal protein intake | At Month 0, 1, 2, and 3
  Via food diaries the total protein intake was calculated
Serum albumin levels | At Month 0, 1, 2, and 3
  throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Susan Sun, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Riverside Medical Center, Riverside, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeloka TK, Dharmatti G, Jamdade T, Pandit M. Are oral protein supplements helpful in the management of malnutrition in dialysis patients? Indian J Nephrol. 2013 Jan;23(1):1-4. doi: 10.4103/0971-4065.107185. PMID 23580797
- [Background] Cano N, Fiaccadori E, Tesinsky P, Toigo G, Druml W; DGEM (German Society for Nutritional Medicine); Kuhlmann M, Mann H, Horl WH; ESPEN (European Society for Parenteral and Enteral Nutrition). ESPEN Guidelines on Enteral Nutrition: Adult renal failure. Clin Nutr. 2006 Apr;25(2):295-310. doi: 10.1016/j.clnu.2006.01.023. Epub 2006 May 12. PMID 16697495
- [Background] Clinical practice guidelines for nutrition in chronic renal failure. K/DOQI, National Kidney Foundation. Am J Kidney Dis. 2000 Jun;35(6 Suppl 2):S17-S104. doi: 10.1053/ajkd.2000.v35.aajkd03517. No abstract available. PMID 10895784